CLINICAL TRIAL: NCT03166423
Title: Clinical Trial Phase I-II of Efficacy and Safety of Snail Slime and Natural Extracts for Healing in Diabetic Foot Ulcers
Brief Title: Efficacy and Safety of Snail Slime and Natural Extracts for Healing in Diabetic Foot Ulcers
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Luis Quiñones Sepulveda, Dr., University of Chile
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CQF-EC-002-14
Record Dates: First submitted 2017-04-24; First posted 2017-05-25 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MU001 patches (Investigational) (Experimental): Patches MU001 (snail slime, calendula extract and propolis extract) more standard of care. Two or three application for week. Treatment until 60 days.
  Patches MU001 (snail slime, calendula extract and propolis extract) on health zone. Three days of treatment.
  Interventions: Drug: MU001 patches (Investigational)
- Conventional patches (Control) (Experimental): Conventional patches approved for diabetic foot ulcers more standard of care. Two or three application for week. Treatment until 60 days.
  Interventions: Device: Conventional patches (Control)

INTERVENTIONS:
Drug: MU001 patches (Investigational) — Patches containing snail slime, calendula extract and propolis extract
  Other Names: MU001 patches
  Arms: MU001 patches (Investigational)
Device: Conventional patches (Control) — Patches containing conventional formulations in medical devices for ulcers (hydrocolloids, activated charcoal silver, alginate, carboxymethylcellulose or hydrogel).
  Other Names: Conventional patches for diabetic foot ulcers
  Arms: Conventional patches (Control)

SUMMARY:
The primary objective is to evaluate the efficacy and safety of the use of a formulation of snail slime and natural extracts, for the curative treatment of ulcer wonds in diabetic foot.

The secondary objetives:

1. To evaluate the efficacy of the use of a formulation of snail slime Helix aspersa Müller and natural extracts (MU001) for the curative treatment of ulcer wonds in diabetic foot with respect to the standard of care, by means the application of patchs that containing the formulation in a treatment period of until 60 days.
2. To determine the safety of the use of a formulation of snail slime Helix aspersa Müller and natural extracts (MU001) in diabetic individuals in a treatment period of until 60 days.

DETAILED DESCRIPTION:
Clinical Study of phase I-II, controlled, simple blind (in relation with biostatistical analysis), randomized, of formulation that containing snail slime Helix aspersa Müller (Cryptophalus aspersus), natural calendula extract, propolis and excipients (MU001).

The formulation in study MU001 wil be added to the standard of care for healing in diabetic foot indicated. The period of recruitment estimated will be 4 month and the follow-up of the patients will be of until 60 days.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes type 2
* Unilateral ulcers
* Grade 1 or grade 2 Wagner ulcers.
* Without infection (except onychomycosis)
* Network family, hygiene, adherence and compliance appropiated

Exclusion Criteria:

* Bilateral ulcers
* Medical conditions with high risk (cancer, allergies)
* Consum of abuse drugs

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2015-11-12 (Actual); Primary Completion 2017-06-01 (Estimated); Study Completion 2017-07-01 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of healing until 60 days or less | 60 days
  Incidence of healing measured with Wagner ulcer classification

SECONDARY OUTCOMES:
Time to healing until 60 days or less | 60 days
  Time to healing measured with Wagner ulcer classification
Incidence of treatment-emergent adverse events (Safety and Tolerability) of a formulation of snail slime and natural extracts in healthy skin | 3 days
  Numbers and types of adverse events in healthy skin of subjects treated with investigational formulation (MU001)
Incidence of treatment-emergent adverse events (Safety and Tolerability) of a formulation of snail slime and natural extracts in ulcer wounds in diabetics foot | 60 days
  Numbers and types of adverse events in ulcers of subjects treated with investigational formulation (MU001)

CONTACTS AND LOCATIONS:
Overall Officials: Luis A. Quiñones Sepúlveda, Dr., Principal Investigator — University of Chile
Locations (4):
- Chile (4):
  - Dirección de salud San Bernardo, Santiago
  - Dirección de Salud El Bosque, Santiago
  - Dirección de salud Independencia, Santiago
  - Dirección de salud San Miguel, Santiago

IPD SHARING:
Plan to Share IPD: No